CLINICAL TRIAL: NCT03741686
Title: Beneficial Effects of Viscous Dietary Fiber From Konjac-Mannan in Subjects With the Insulin Resistance Syndrome
Brief Title: Effect of Konjac-mannan in Individuals With Insulin-Resistance Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Dicofarm (Other); University of Toronto, Toronto (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Konjac in Insulin Resistance
Record Dates: First submitted 2018-11-07; First posted 2018-11-15 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Insulin Resistance Syndrome
Keywords: insulin resistance syndrome; fiber; konjac
MeSH Terms: conditions — Metabolic Syndrome | interventions — (1-6)-alpha-glucomannan; Dietary Fiber

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Konjac-mannan (Experimental): Konjac-mannan fiber-enriched biscuits with NCEP Step II metabolically controlled diet.
  Interventions: Dietary Supplement: konjac glucomannan
- Placebo (Placebo Comparator): wheat bran fiber biscuits with NCEP Step II metabolically controlled diet.
  Interventions: Dietary Supplement: wheat bran

INTERVENTIONS:
Dietary Supplement: konjac glucomannan — Konjac-mannan fiber-enriched biscuits (0.5 g/412KJ [100kcal] of glucommanan)
  Arms: Konjac-mannan
Dietary Supplement: wheat bran — Wheat bran (hard red wheat bran) fiber enriched biscuits
  Arms: Placebo

SUMMARY:
To study whether a diet high in fiber from Konjac-mannan (KJM) has an effect on metabolic control in individuals with insulin resistance syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Impaired glucose tolerant
* Clinical absent of CHD
* BMI less than 30 kg/m2
* Presence of full insulin resistance syndrome
* Reduced HDL cholesterol
* Elevated serum triglycerides
* Moderate hypertension

Exclusion Criteria:

* Regular smoking
* Regular alcohol consumption
* Family history of premature coronary heart disease
* Hypothyroidism
* Renal, hepatic or gastrointestinal disease
* Taking medications for hyperglycemia
* Taking medications for hyperlipidemia
* Taking medications for hypertension

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 1991-01 (Actual); Primary Completion 1992-06 (Actual); Study Completion 1999-06 (Actual)

PRIMARY OUTCOMES:
change in total:HDL cholesterol | change from baseline after 3 weeks, relative to control
change in fructosamine | change from baseline after 3 weeks, relative to control
change in systolic blood pressure | change from baseline after 3 weeks, relative to control

SECONDARY OUTCOMES:
change in total cholesterol | change from baseline after 3 weeks, relative to control
change in LDL cholesterol | change from baseline after 3 weeks, relative to control
change in HDL cholesterol | change from baseline after 3 weeks, relative to control
change in apolipoprotein A-1 | change from baseline after 3 weeks, relative to control
change in apolipoprotain B | change from baseline after 3 weeks, relative to control
change in glucose | change from baseline after 3 weeks, relative to control
change in insulin | change from baseline after 3 weeks, relative to control
change in diastolic blood pressure | change from baseline after 3 weeks, relative to control
change in body weight | change from baseline after 3 weeks, relative to control
change in apoB:ApoA-1 | change from baseline after 3 weeks, relative to control